CLINICAL TRIAL: NCT01789125
Title: Augmenting Smoking Cessation With Transdiagnostic CBT for Smokers With Anxiety
Brief Title: Smoking Termination / Anxiety Reduction Treatment (ST/ART)
Acronym: START
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Michael J. Zvolensky, Ph.D., Hugh Roy and Lillie Cranz Cullen Distinguished University Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34DA03131301A1; R34DA031313 (NIH)
Record Dates: First submitted 2013-02-08; First posted 2013-02-11 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Smoking; Anxiety Disorders
Keywords: anxiety; stress; smoking; cessation
MeSH Terms: conditions — Smoking; Anxiety Disorders | interventions — Tobacco Use Cessation Devices; Transdermal Patch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Smoking Termination and Anxiety Reduction Treatment (Active Comparator): Cognitive-behavioral treatment program that blends smoking cessation and anxiety reduction treatment strategies
  Interventions: Drug: Nicotine Patch; Behavioral: Smoking Termination and Anxiety Reduction Treatment
- Educational-Support Psychotherapy (Active Comparator): Educational-based psychotherapy and standard smoking cessation treatment program
  Interventions: Drug: Nicotine Patch; Behavioral: Education-Supportive Psychotherapy

INTERVENTIONS:
Drug: Nicotine Patch
  Other Names: Patch; NRT
Behavioral: Smoking Termination and Anxiety Reduction Treatment — Integrated smoking cessation and anxiety reduction treatment
  Arms: Smoking Termination and Anxiety Reduction Treatment
Behavioral: Education-Supportive Psychotherapy
  Arms: Educational-Support Psychotherapy

SUMMARY:
The primary aim of this research study is to enhance smoking cessation outcome among smokers with anxiety disorders. The investigators are comparing two group treatment approaches: (1) An educational-supportive psychotherapy and standard smoking cessation treatment, and (2) An integrated smoking cessation and anxiety treatment program (START). Both treatments also utilize nicotine replacement therapy.

DETAILED DESCRIPTION:
The chief objective of the proposed study is to develop an integrated standard smoking cessation treatment and transdiagnostic anxiety disorder treatment for smokers with anxiety disorders. The intervention is designed to promote smoking cessation and reduce (a) anxiety symptoms, (b) depression, and (c) the cognitive factor of AS, thereby reducing three notable emotional risk factors of smoking cessation relapse, while at the same time targeting (d) nicotine withdrawal symptoms. The intervention development approach will follow a staged model consistent with NIH guidelines for developing and standardizing behavioral therapies. During the first year, startup activities will include piloting the integrated intervention on a subset of individuals, soliciting internal and external expert consultant and participant feedback, and development of the final treatment protocol. The goal during this phase of the project will be to establish feasibility of treatment delivery, participant acceptability, and potential for an effect. During the following two years, a pilot two-arm efficacy study will be undertaken. The two arms of the randomized trial (RCT) will be: (a) the integrated smoking cessation treatment, consisting of a standard smoking cessation intervention (i.e., CBT-Smoking + Nicotine Replacement Therapy [NRT]) plus a transdiagnostic CBT for anxiety (Smoking Termination and Anxiety Reduction Treatment; START) or (b) standard smoking cessation intervention (i.e., CBT-Smoking + NRT) plus contact control (ST+CTRL). The primary outcomes will be short- and long-term point prevalence abstinence (PPA) and time to first smoking lapse and relapse. The following specific aims are proposed: 1. To compare, in a pilot RCT, the effects of START vs. ST+CTRL on smoking cessation outcomes: Short- and longterm PPA. The investigators expect that PPA will be higher, both in the short- and longterm, for those in the START condition compared to those in ST+CTRL. Similarly, The investigators expect the rate of decline in abstinence over time to be slower in START than in ST+CTRL Time to first smoking lapse and time to smoking relapse. The investigators expect mean time to first lapse and to relapse to be greater for those in the START compared to those in the ST+CTRL condition. 2. To compare, in a pilot RCT, the effect of START vs. ST+CTRL on the remission of anxiety disorders, anxiety and depressive symptoms, anxiety sensitivity, and nicotine withdrawal symptoms. 3. To explore the mechanisms by which START improves smoking cessation. The investigators expect that: Treatments over time will directly cause changes in abstinence and withdrawal symptoms, AS, anxiety symptoms, depressed mood (i.e., the proposed mediators of change in abstinence); The effect of treatment on anxiety symptoms and depressed mood will be moderated by treatment condition, such that those receiving START will improve more than those receiving ST+CTRL Changes in each mediator over time will lead to improvements in abstinence over time, and decreases in AS over time will lead to improvements in anxiety symptoms and depressed mood over time.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65 years old
* Capable of providing informed consent
* Willing to attend all study visits and comply with the protocol
* Daily smoker for at least one year
* Currently smoke an average of at least 6 cigarettes per day
* Report a motivation to quit smoking in the next 6 weeks of at least 5 on a 10-point scale

Exclusion Criteria:

* Use of other tobacco products
* Current or past psychotic disorders of any type, or comorbid psychiatric conditions that are relative or absolute contraindications to the use of any treatment option in the study protocol
* Currently suicidal or high suicide risk
* Current use of any pharmacotherapy or psychotherapy for smoking cessation not provided by the researchers during the quit attempt
* Unwilling to cease use of benzodiazepines or other fast-acting anxiolytics
* Concurrent psychotherapy initiated in the past three months, or ongoing anxiety psychotherapy
* Current or intended participation in a concurrent substance abuse treatment
* Insufficient command of English to participate in assessment or treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Short- and long-term point prevalence abstinence | Change from baseline at 1, 2, 4, 8, 10, 16, and 24 weeks post quit day.
  The investigators will ask participants various questions about their abstinence. The investigators will measure the length of time between when treatment ends and when/ if they start smoking again. The unit of measure will be length of time in days.

SECONDARY OUTCOMES:
Time to first smoking lapse and relapse | Change from baseline at 1, 2, 4, 8, 10, 16, and 24 weeks post quit day.
  The investigators will ask participants to record the time (in days) of their first (if any) lapse in smoking and their relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Zvolensky, Ph.D., Principal Investigator — University of Houston
Locations (1):
- Anxiety and Health Research Laboratory and Substance Use Treatment Clinic, University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Data will be made available upon request.